CLINICAL TRIAL: NCT05353036
Title: Expanded Preoperative Survey During Perioperative Care to Identify Substance Use in Teenagers and Adolescents
Brief Title: Survey to Identify Substance Use in Teenagers and Adolescents
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: STUDY00002306
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents: Patients 12-21 years undergoing anesthetic care
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey assessing incidence, frequency, and type of illicit substance use

SUMMARY:
This is a prospective survey study of patients 12-21 years undergoing anesthetic care. The primary objective is to determine the incidence of illicit substance use and abuse prior to anesthetic care. The secondary objective is to determine the illicit substances used and their frequency in patients presenting for anesthetic care.

DETAILED DESCRIPTION:
The participants will be asked to complete a survey in REDCap using an iPad during the visit. The study will record any positive answers from the drug and tobacco use questions routinely asked of the parents during the on-line pre-admission testing process. These include yes/no answers regarding drug, alcohol, and tobacco use.

The information collected will include only demographic data including age, weight, gender, ethnicity/race, and zip code. Survey data will be coded and will not include patient information. Completion of the survey will take approximately 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 12-21 years of age
* Presenting for surgery or procedure requiring anesthesia

Exclusion Criteria:

* Patients who are not able to complete the computerized survey due to physical or intellectual impairment
* Patients who are non-English speaking

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents undergoing procedure requiring anesthesia at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Adolescents: Patients 12-21 years undergoing anesthetic care
  Survey: REDCap survey assessing incidence, frequency, and type of illicit substance use
Period: Overall Study
Arm/Group | Adolescents
Started | 250
Completed | 250
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adolescents
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 109
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 37
  White | 187
  More than one race | 12
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 250

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adolescent and Parent Reported Alcohol, Drug, Vaping and Tobacco Usage
Description: As part of standard of care, nurses contact the parents of children scheduled for surgery to obtain health history and any alcohol, drug, vaping and tobacco usage. For the study, adolescents were asked to complete a survey on REDCap regarding their alcohol, drug, vaping and tobacco usage and those responses were compared to the answers the parents gave to the nurses during pre-op phone call.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Total responses from both participants and parents.
- Adolescents: Patients 12-21 years undergoing anesthetic care
  Survey: Survey assessing incidence, frequency, and type of illicit substance use via REDCap
- Parents: Parents of the adolescent participants
Arm/Group | Overall | Adolescents | Parents
Number analyzed (Participants) | 500 | 250 | 250
Participants
  Alcohol: No response recorded | 1 | 1 | 0
  Alcohol: No | 425 | 180 | 245
  Alcohol: Yes | 74 | 69 | 5
  Drug use: No | 437 | 198 | 239
  Drug use: Yes | 63 | 52 | 11
  Vaping: No response recorded | 1 | 1 | 0
  Vaping: No | 448 | 209 | 239
  Vaping: Yes | 51 | 40 | 11
  Tobacco: No response recorded | 1 | 1 | 0
  Tobacco: No | 482 | 237 | 245
  Tobacco: Yes | 17 | 12 | 5

2. Primary Outcome: Alcohol Use
Description: Adolescents were asked in a REDCap survey Do you currently or have you ever drank alcohol?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 250
Participants
  No response recorded | 1
  No | 180
  Yes | 69

3. Primary Outcome: Marijuana Use
Description: Adolescents were asked in a REDCap survey Do you currently or have you ever smoked or consumed marijuana, THC, or cannabis?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 250
Participants
  No response recorded | 1
  No | 198
  Yes | 51

4. Primary Outcome: Vape Pen Use
Description: Adolescents were asked in a REDCap survey Do you currently or have you ever vaped?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 250
Participants
  No response recorded | 1
  No | 209
  Yes | 40

5. Primary Outcome: Tobacco Use
Description: Adolescents were asked in a REDCap survey Do you currently or have you ever used tobacco?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 250
Participants
  No response recorded | 1
  No | 237
  Yes | 12

6. Primary Outcome: Prescription Opioid Use for Acute Pain
Description: Adolescents were asked in a REDCap survey Do you currently or have you ever used a prescribed opioid for acute pain?
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 250
Participants
  No | 215
  Yes | 35

7. Secondary Outcome: Most Recent Alcohol Use
Description: Adolescents were asked in a REDCap survey When was the last time you used alcohol?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used alcohol question.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 69
Participants
  Not currently using | 15
  Within the last 24 hours | 2
  Within the last week | 11
  Within the last year | 41

8. Secondary Outcome: Age First Drank Alcohol
Description: Adolescents were asked in a REDCap survey How old were you when you first drank alcohol?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever drank alcohol question.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Adolescents
Number analyzed (Participants) | 69
years | 16 [14 to 17]

9. Secondary Outcome: Most Recent Marijuana Use
Description: Adolescents were asked in a REDCap survey When was the last time you used marijuana?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used marijuana question.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 51
Participants
  Not currently using | 10
  Within the last 24 hours | 6
  Within the last week | 16
  Within the last year | 19

10. Secondary Outcome: Age First Used Marijuana
Description: Adolescents were asked in a REDCap survey How old were you when you first started using?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used marijuana question.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Adolescents
Number analyzed (Participants) | 51
years | 16 [14 to 17]

11. Secondary Outcome: Most Recent Vape Pen Use
Description: Adolescents were asked in a REDCap survey When was the last time you vaped?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used vape pen question.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 40
Participants
  Not currently using | 11
  Within the last 24 hours | 10
  Within the last week | 12
  Within the last year | 7

12. Secondary Outcome: Age First Started Vaping
Description: Adolescents were asked in a REDCap survey How old were you when you first started vaping?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever vaped question.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Adolescents
Number analyzed (Participants) | 40
years | 15.5 [14 to 16]

13. Secondary Outcome: Most Recent Tobacco Use
Description: Adolescents were asked in a REDCap survey When was the last time you used tobacco?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used tobacco question.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 12
Participants
  Not currently using | 5
  Within the last 24 hours | 3
  Within the last week | 2
  Within the last year | 2

14. Secondary Outcome: Age First Used Tobacco
Description: Adolescents were asked in a REDCap survey How old were you when you started using tobacco?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used tobacco question.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Adolescents
Number analyzed (Participants) | 12
years | 15 [14 to 15.5]

15. Secondary Outcome: Most Recent Prescribed Opioid Use
Description: Adolescents were asked in a REDCap survey When was the last time you used a prescribed opioid for acute pain?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or have ever used a prescribed opioid for acute pain question.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 35
Participants
  Not currently using | 13
  Within the last 24 hours | 3
  Within the last week | 3
  Within the last year | 15
  No answer | 1

16. Secondary Outcome: Prescribed Opioid Use for Anything Other Than Pain
Description: Adolescents were asked in a REDCap survey Did you ever use that medication (prescribed opioid) for anything other than pain?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used prescribed opioid for acute pain question.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 35
Participants
  No | 33
  Yes | 2

17. Secondary Outcome: Prescribed Opioid Use Leading to Abuse
Description: Adolescents were asked in a REDCap survey Did your using prescribed opioid for anything other than pain lead to your abusing opioids/narcotics?
Time Frame: Baseline
Population: The number of participants that answered yes to the currently or ever used prescribed opioid for acute pain question.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents
Number analyzed (Participants) | 35
Participants
  No | 34
  Yes | 1

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Adolescents
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 0/250

LIMITATIONS AND CAVEATS:
One of the limitations of this study is the fact that data were only collected during the summer months. It is possible that these data would differ if collected throughout the school year. Additionally, the surveys were collected from patients undergoing prescheduled surgical procedures. Due to the rapid nature of urgent or emergent cases, inclusion of these patients in the study cohort was not deemed feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT05353036/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT05353036/SAP_001.pdf